CLINICAL TRIAL: NCT07020754
Title: Effect of Arginine- and Glutamine-based Oral Formulations on Salivary Biomarkers and Clinical Severity of Radiation-induced Oral Mucositis in Head and Neck Cancer: A Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma ElSayed, assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUE.REC25/8-2025
Record Dates: First submitted 2025-06-06; First posted 2025-06-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Radiation Induced Oral Mucositis; Oral Mucositis; Oral Mucositis Due to Radiation
Keywords: Radiation-induced oral mucositis (RIOM); Head and neck cancer (HNC); L-arginine; Epidermal growth factor (EGF); L-glutamine
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I - L-arginine + Maltodextrin Oral Suspension (Experimental): Patients receive 5 g of L-arginine + 5 g of maltodextrin dissolved in cold distilled water.
  Interventions: Dietary Supplement: L-arginine Oral Suspension
- Group II - Glutamine + Maltodextrin Oral Suspension (Active Comparator): Group II - Glutamine + Maltodextrin Oral Suspension
  Interventions: Dietary Supplement: L-glutamine Oral Suspension
- Group III - Maltodextrin Oral Suspension (Control Group) (Placebo Comparator): Patients receive 10 g of maltodextrin only, prepared and administered identically to the other groups.
  Interventions: Dietary Supplement: Maltodextrin Oral Suspension (Control)

INTERVENTIONS:
Dietary Supplement: L-arginine Oral Suspension — Type: Dietary supplement
  Dosage: 5 g L-arginine + 5 g maltodextrin
  Route: Oral (swish-and-swallow)
  Frequency: Three times daily, 30 minutes before meals
  Duration: From the 2nd to the 7th week of radiotherapy
  Arms: Group I - L-arginine + Maltodextrin Oral Suspension
Dietary Supplement: L-glutamine Oral Suspension — Type: Dietary supplement
  Dosage: 5 g L-glutamine + 5 g maltodextrin
  Route: Oral (swish-and-swallow)
  Frequency: Three times daily, 30 minutes before meals
  Duration: From the 2nd to the 7th week of radiotherapy
  Arms: Group II - Glutamine + Maltodextrin Oral Suspension
Dietary Supplement: Maltodextrin Oral Suspension (Control) — Type: Placebo comparator
  Dosage: 10 g maltodextrin
  Route: Oral (swish-and-swallow)
  Frequency: Three times daily, 30 minutes before meals
  Duration: From the 2nd to the 7th week of radiotherapy
  Arms: Group III - Maltodextrin Oral Suspension (Control Group)

SUMMARY:
This triple-blinded, randomized controlled clinical trial investigates the effectiveness of L-arginine and L-glutamine oral suspensions in managing radiation-induced oral mucositis (RIOM) in patients with head and neck cancer (HNC) undergoing radiotherapy. A total of 69 patients are randomly assigned to three groups: L-arginine + maltodextrin, glutamine + maltodextrin, or maltodextrin alone (control).

The interventions are administered as a swish-and-swallow solution three times daily from the second to seventh week of radiotherapy. Key outcomes assessed include oral mucositis severity (WHO scale), pain intensity (VAS), body mass index (BMI), oral health-related quality of life (OHIP-14), and salivary epidermal growth factor (EGF) levels. The study aims to determine whether L-arginine offers superior mucosal healing and symptom relief compared to glutamine or placebo.

DETAILED DESCRIPTION:
Radiation-induced oral mucositis (RIOM) is recognized as a frequent and severe complication among patients with head and neck cancer (HNC) who undergo radiotherapy (RT) 1. It manifests as damage to healthy tissues, specifically inflammation and/or ulceration of the oral mucosa, affecting over 80% of these patients receiving radiation therapy 2.

RIOM manifests as a normal tissue injury lasting from 7 to 98 days, initiated by acute inflammation in the oral mucosa, tongue, and pharynx following RT exposure 1. This inflammation is accompanied by the accumulation of various inflammatory cells and the secretion of cytokines, chemotactic agents, and growth factors. RIOM may escalate into a life-threatening condition due to significant blockages that restrict the intake of food and water, leading to weight loss and septic issues from the loss of protective epithelial and basement membrane layers. Consequently, these complications can disrupt cancer treatment and necessitate changes in the radiation dose, thus impacting local tumor control.3 The pathogenesis of RIOM associated with RT for HNC unfolds through a complex, multi-stage process. Initially, ionizing radiation directly damages cellular DNA within the radiation field, resulting in lethal double-strand breaks. When these breaks are not repaired accurately, it leads to programmed cell death or apoptosis. Concurrently, this radiation exposure stimulates various cells such as endothelial cells and fibroblasts to produce reactive oxygen species (ROS). These ROS further exacerbate DNA damage and disrupt cellular functions by modifying protein and lipid membrane structures, leading to escalated inflammation 4.

When excessive ROS accumulate, they cause oxidative stress, managed by antioxidants like superoxide dismutase and glutathione peroxidase. Disruptions in this balance lead to oxidative damage, increasing the risk of cancer and inflammatory conditions. Chemoradiation activates NF-kappa B, heightening pro-inflammatory cytokine levels that drive the progression to mucosal ulceration characteristic of OM. This condition severely impacts patients' nutrition and oral hygiene and increases the risk of secondary infections due to deeper tissue damage 5.

L- glutamine is L-alpha-amino acid. It is the most abundant free amino acid in human blood. L- glutamine is needed for several functions in the body including for the synthesis of proteins as well as an energy source. L-glutamine can be synthesized by the body and can also be obtained from the diet if needed.6 L- glutamine is crucial for powering lymphocytes and the gastrointestinal tract, helping to protect against infections and maintaining the mucosal barrier. It's important in cellular metabolism and acts as a nitrogen carrier across various tissues. Although its plasma levels remain stable, glutamine is predominantly stored in muscles and regulated by the liver 7. Several studies indicated that glutamine could decrease both the frequency and intensity of OM 8-13.

L-arginine, a conditionally essential amino acid, is primarily metabolized by enzymes such as nitric oxide synthase (NOS), arginine decarboxylase, and arginase (ARG), contributing to the synthesis of proteins and various bioactive molecules like nitric oxide (NO), proline, creatine, and polyamines 14. There is growing interest in enhancing the physiological roles of arginine, particularly in reducing intestinal inflammation and oxidative stress 15. Previous research has shown that L-arginine supplementation in both animals and humans with intestinal disorders can lessen intestinal damage, alleviate oxidative stress and inflammation, and help reestablish mucosal immune balance. Notably, Coburn et al. have documented that L-arginine supplementation reduced intestinal inflammation in mouse models of dextran sulfate sodium (DSS)- induced colitis, an experimental model of IBD.16 L-arginine significantly enhances wound healing through various mechanisms. It is crucial for collagen synthesis, which is fundamental for new tissue development and the formation of strong connective tissue. This amino acid also has anti-inflammatory effects that regulate the body's response to injury, reducing the risk of chronic inflammation that can impede healing. Additionally, l-arginine promotes fibroblast proliferation, which is essential for producing collagen and other extracellular matrix components that aid in wound repair. Indirect benefits of l-arginine include improved circulation and blood flow to the wound area, supplying necessary oxygen and nutrients, and bolstering the immune system to fight infections and support healing processes 17-20.

Based on the various physiological properties of L-arginine, its anti-inflammatory effects, and its capacity for wound healing and tissue repair, this study aim to evaluate the effect of L-arginine oral suspension versus glutamine oral suspension on salivary EGF, and on management of radiation-induced oral mucositis (RIOM) and its associated symptoms, as well as assessing their effects on the oral health related quality of life in HNC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 70 years

Diagnosed with head and neck cancer (HNC) and undergoing radiotherapy (RT)

Development of oral mucositis during the 2nd to 3rd week of RT

Receiving a minimum radiation dose of 50 Gy to the oral cavity

Undergoing intensity-modulated radiotherapy (IMRT) with three-dimensional conformal techniques after complete tumor resection

Ability and willingness to provide informed consent

Able to comply with study procedures and follow-up assessments

Exclusion Criteria:

* History of prior radiotherapy

Diagnosed with diabetes mellitus

Presence of salivary gland tumors

Renal or hepatic insufficiency

Sepsis or any active systemic infection

Distant metastases

Any condition that may interfere with oral sample collection or affect EGF levels (e.g., autoimmune oral disease)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-25 (Actual)

PRIMARY OUTCOMES:
Change in salivary IL-6 levels during radiotherapy-induced oral mucositis | From week 2 of radiotherapy (baseline) , week 5 of radiotherapy (peak mucositis phase, week 7 of RT
  Salivary interleukin-6 (IL-6) concentration will be measured using enzyme-linked immunosorbent assay (ELISA) to assess inflammatory response during radiotherapy. The primary endpoint is the between-group difference in IL-6 change from baseline to peak mucositis following arginine-, glutamine-, or maltodextrin-based oral intervention. IL-6 was selected as the primary biomarker due to its established role in radiation-induced oral mucosal inflammation and association with mucositis severity.

SECONDARY OUTCOMES:
Change in Salivary Epidermal Growth Factor (EGF) Levels | Baseline (2nd week of radiotherapy), week 5 of radiotherapy (peak mucositis phase) End of treatment (7th week)
  Description:
  Measures the concentration of salivary EGF, a key biomarker involved in mucosal healing and epithelial regeneration. This outcome assesses whether L-arginine or L-glutamine can enhance EGF production, contributing to faster recovery from oral mucositis.
  Method:
  Whole saliva is collected under stimulation, processed, and analyzed using ELISA (Enzyme-Linked Immunosorbent Assay).
Change in salivary nitric oxide levels during radiotherapy-induced oral mucositis | From week 2 of radiotherapy (baseline) to week 5 (peak mucositis) and week 7 (end of radiotherapy)
  Salivary nitric oxide concentration, expressed as total nitrite/nitrate levels, will be quantified using a colorimetric assay to evaluate oxidative and inflammatory signaling during radiotherapy. The outcome measure is the between-group difference in nitric oxide change from baseline to peak mucositis and end of radiotherapy following arginine-, glutamine-, or maltodextrin-based oral intervention. Nitric oxide is included as a secondary biomarker due to its dual role in radiation-induced oxidative stress and mucosal wound healing.
Severity of Oral Mucositis | 2nd, 5th, and 7th weeks of radiotherapy
  Assessed using the WHO Oral Toxicity Scale, which grades mucositis from 0 (no symptoms) to 4 (severe ulceration requiring feeding support). This measure reflects the extent of mucosal injury caused by radiotherapy and the potential protective effect of interventions.
Pain Intensity | 2nd, 5th, and 7th weeks of radiotherapy
  Evaluated using the Visual Analogue Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain). This subjective measure tracks changes in patient-reported pain severity throughout treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Future University in Egypt, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided